CLINICAL TRIAL: NCT02770534
Title: Assessing the Utility of Thromboelastography (TEG) and Endogenous Thrombin Potential (ETP) in Adults With Sickle Cell Disease
Brief Title: Evaluating Thromboelastography (TEG) and ETP in Sickle Adults
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GuysThomasNHS
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Sickle patients in steady state: Well sickle cell patients attending the outpatient clinic
  Interventions: Procedure: blood test
- Sickle cell patients admitted in crisis: Inpatients with acute vaso-occlusive crisis
  Interventions: Procedure: blood test
- Sickle patients on transfusion program: Sickle patients managed on a regualar transfusion program
  Interventions: Procedure: blood test
- Sickle patients on Hydroxycarbamide: Sickle cell patients managed on hydroxycarbamide and on a stable dose for at least 3 months
  Interventions: Procedure: blood test
- Health controls: Well age and race matched individuals without a known diagnosis of sickle cell anaemia
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: blood test — 10mls extra mls of blood taken during usual phlebotomy procedures

SUMMARY:
The primary aim of this study is to investigate the reported enhanced coagulation status (prothrombotic status) in patients with sickle cell disease using 2 laboratory tests; thromboelastography (TEG) and Endogenous Thrombin Potential (ETP), and comparing the results to healthy race matched controls to ascertain if there is a significant difference. Race matching of the control participants is being carried out due to the well reported racial differences in coagulation parameters that exist in healthy individuals. The investigators are aiming to study the clotting state in sickle patients on regular transfusion therapy and those on hydroxycarbamide, both treatments offered to sickle patients to ameliorate the condition. The study will assess the reported prothrombotic state using TEG and ETP.

DETAILED DESCRIPTION:
Sickel cell disease (SCD) is the most common inherited red cell disorder worldwide, the genetic mutation in SCD results in the production of abnormal haemoglobin (HbS). This leads to anaemia and unpredictable painful episodes referred to as a sickle cell crisis. Sickle cell crises result in significant chronic health problems including stroke, kidney failure, breathing problems, leg ulcers and chronic and ultimately leads to a decrease in life expectancy.

The method by which sickling results in the above issues is recognised as very complex and it is thought these patients may have enhanced blood clotting which may play a role in the complications they get. Sickle cell patients are reported to have higher risk of blood clots such as deep vein thrombosis.

The primary aim in this study is to investigate the reported enhanced coagulation status in sickle cell adult sickle cell patients using 2 laboratory tests, thromboelastography (TEG) and Endogenous Thrombin Potential (ETP) , the investigators will compare the results in sickle participants to healthy race matched control participants to show if there is a significant difference. The investigators also aim to study the coagulation status in sickle participants on a variety of treatments such as transfusion and hydroxycarbamide, both treatments offered to sickle patients. Many trials have shown the benefits of both transfusions and hydroxycarbamide in SCD, they reduce the risk of stroke and frequency with which patients get crises.

To the best of teh investigators knowledge this will be the first study evaluating the clinical utility of TEG and ETP in adult patients with SCD

The trial will be conducted in compliance with the principles of the Declaration of Helsinki and the principles of Good Clinical Practice. It has been submitted for approval to the London NHS Research Ethics Committee.

Trial Design & Flowchart This is a cross sectional case controlled clinical study in patients with sickle cell disease. Control participants will be race and age matched participants without sickle cell disease. Written informed consent will be obtained from all participants. The samples will be taken as part of the usual clinic or inpatient procedure with 10 extra millilitres of blood venesected at a phlebotomist or nurse scheduled to venesect participants as part of their usual medical care. Healthy controls will be asked to provide a 10ml blood sample which will be taken by a qualified member of staff. The investigators are aiming to collect samples from 100 patients in total and 20 healthy controls for comparison

ELIGIBILITY:
Inclusion Criteria: Patient participants must be over 16 years of age with sickle disease HbSS or HbSb0, SCD genotype which must have been previously confirmed by high performance liquid chromatography with results on GSTT trust electronic patient record (EPR), all participants must be able to give written consent.

Exclusion Criteria:

currently pregnant have a known diagnosis of an inherited bleeding disorder such as e.g. von willebrand disease on anticoagulant therapy, have severe liver disease with liver transaminases greater than 5x upper limit of normal.

Healthy control paticipants will be race and age matched to the patient cohort and must also not be currently pregnant, have a known diagnosis of an inherited bleeding disorder such as e.g. von willebrand disease. The investigators will also exclude healthy participants on anticoagulant therapy as well as those with severe liver disease and liver transaminases greater than 5x upper limit of normal.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult sickle cell patients ( age 16+)attending registered and attending the service at Guys adn St Thomas Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
results of TEG and ETP analysis:results confirming enhanced coagulation state in sickle cell patients | 4 months
  completions of analysis of all subjects and controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No